CLINICAL TRIAL: NCT03285191
Title: Patient Interviews to Better Understand Disease Experience and Unmet Treatment Needs in Rheumatoid Arthritis
Brief Title: Subject Insights to Understand Rheumatoid Arthritis (RA)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 206577
Record Dates: First submitted 2017-06-29; First posted 2017-09-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Arthritis, Rheumatoid
Keywords: NRS; Concept elicitation; Real-time data capture; Rheumatoid arthritis; GSK3196165
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects participating in the CE interview: Thirty subjects (comprised of n=15 csDMARD-IR and n=15 bDMARD-IR) will participate in the CE interview.
  Interventions: Other: Numerical rating scale
- Subjects participating in interview and real-time data capture: Ten of the thirty CE interview participants will be offered the opportunity to participate in the real-time data capture App substudy.
  Interventions: Other: Numerical rating scale; Other: Real-time data capture app

INTERVENTIONS:
Other: Numerical rating scale — Following the concept elicitation interview, participants will be presented with a list of typical RA symptoms and asked to rank how bothersome each symptom is and how important it would be to improve with treatment on a 1-5 numerical rating scale (NRS).
Other: Real-time data capture app — Real time data capture app is a smart-phone or web-based application which will allow the subjects to provide responses about their experience of HOA in real-time via varying video, audio, photographic and text forms using a study-specific application on their own smart device. Up to ten of the thirty interview participants can participate in the app sub study, which is voluntary.
  Groups: Subjects participating in interview and real-time data capture

SUMMARY:
Rheumatoid arthritis (RA) is a chronic, systemic autoimmune disease affecting the joints and can lead to joint pain, swelling, redness and stiffness and can cause deformity, loss of strength and immobility. This cross-sectional qualitative study aims to explore the burden of established RA by conducting semi-structured Concept elicitation (CE) interviews (60 minutes duration) and real-time data capture task. The conceptual model developed from this data will be used to support the development of GSK3196165, a recombinant human monoclonal antibody (mAb) targeted for the treatment of RA. The CE interviews will explore the subject experience of RA and will collect information about symptoms, disease impact on functioning and health related quality of life (HRQoL), and treatment experiences/impacts of the condition and the language used by subjects to describe them. Following the CE interview, subjects will be asked to complete a brief symptom ranking exercise where they will need to rank how bothersome each RA symptom is and how important it would be to improve with treatment on a 1-5 numerical rating scale (NRS). After the interviews, the real-time disease experience of subjects will be captured by the real-time data capture app-based activity over a period of 7 days. Approximately 30 English-speaking subjects from the United States (US) with RA who are inadequate responders of conventional synthetic disease-modifying anti-rheumatic drugs (csDMARDs) and/or (bDMARDs) will participate in the interviews and of these, 10 subjects will be offered the opportunity to participate in the real-time data capture sub study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged >=18 years or over.
* Subject has a diagnosis of rheumatoid arthritis and has had this diagnosis for at least 6 months.
* Subject has a minimum of four swollen and tender joints.
* Subject is either an inadequate responder to csDMARDs and has never received a bDMARD or an inadequate responder to bDMARDs (subject may be receiving bDMARDs only or may be continuing csDMARD treatment in addition to receiving a bDMARD).
* Subject is willing and able to participate in the study and provide written informed consent.
* Subject is a fluent US-English speaker and is able to read, write and fully understand the US-English language.
* Subject is willing and able to participate in a 60-minute interview and optional app task to discuss their experience of rheumatoid arthritis.

For subjects taking part in real-time data capture:

* Subject owns/or has access to either a smartphone [iPhone Operating System (iOS) or android] or tablet which has video, audio/microphone and photographic capabilities and access to either the Apple app store or Google play store to download the app.
* Subject is willing and able to take part in the real time data application task and respond to a series of questions/tasks fielded via the application over the course of seven days and is willing to respond to some brief questions following the real-time data capture task about their experience of using the app and completing the tasks, in a 5-10 minute telephone call.
* Subject would feel comfortable recording short videos of themselves and providing audio commentary in response to app questions/tasks.

Exclusion Criteria:

* Subject has a history of other inflammatory rheumatological or autoimmune disorders that are not secondary to RA.
* Subject has significant unstable or uncontrolled acute or chronic disease other than RA.
* Subject is unwilling or unable to comply with the requirements of the study or has a physical or mental condition that, in the opinion of the physician, may affect the subject's ability to participate in the study, the responses he/she might provide or their ability to provide consent.
* Subject is currently or has previously been enrolled in a clinical trial for RA in the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty English speaking subjects from the US with RA who are inadequate responders to csDMARDs and/or bDMARDs will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2017-08-17 (Actual); Study Completion 2017-08-17 (Actual)

PRIMARY OUTCOMES:
Number of subjects with RA participating in CE interviews | 1 day
  CE interviews will be carried out to explore disease experience with respect to symptoms, impacts and treatment/surgical experiences.

SECONDARY OUTCOMES:
Analysis of RA experience by using real-time data data capture task | Up to 7 days
  A subgroup of ten of the thirty subjects participating in the CE interviews will be asked to take part in the real-time data capture task over the course of 7 days and during this time a series of 5-7 questions/tasks will be asked to subjects via the application to explore the experience of the symptoms, HRQoL impacts, treatment of RA and any day-to-day variability that exists in real time'.
Preparation of the conceptual model | Up to 7 days
  Data obtained from the CE interviews and real-time data capture as well as literature reviews will be used to develop a conceptual model for RA. Symptom, impact, and treatment concepts which have been identified will be grouped into domains and displayed visually and any identified relationships or trends between domains will also be included in the model. A contents key will be developed to show the source of the concept.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bollington, Cheshire, United Kingdom

REFERENCES:
- See also: Results for study 206577 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/206577?search=study&study_ids=206577#rs